CLINICAL TRIAL: NCT01679054
Title: Cost-minimization Analysis of Xeloda® vs 5-fluorouracil-based Treatment for Gastric Cancer Patients in Hong Kong
Brief Title: Cost-minimization Analysis of Gastric Cancer Treatments in Hong Kong
Status: Completed | Type: Observational
Sponsor: Vivian Wing Yan Lee (Other)
Collaborators: Hoffmann-La Roche (Industry); Princess Margaret Hospital, Hong Kong (Other Government); Pamela Youde Nethersole Eastern Hospital (Other)
Responsible Party: Sponsor-Investigator, Vivian Wing Yan Lee, Associate Professor, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Other Study IDs: Roche-TR116582; TR116582VLKZ001 (Other: CUHK)
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Results first posted 2024-03-12 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-08

CONDITIONS: Gastric Cancer
Keywords: Neoplasm; Gastric Cancer; Cost
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- EOX: Epirubicin + Oxaliplatin + Capecitabine (EOX) Epirubicin 50 mg/m2 iv bolus d1 q3w x 8 cycles Oxaliplatin (Eloxatin) 130 mg/m2 iv over 2 hours d1 q3w x 8 cycles Capecitabine (Xeloda) 625 mg/m2 po bid x 6 months
- FOLFOX4: FOLFOX4 Leucovorin 200 mg/m2 iv over 2 hrs before 5-FU, d1 and 2 5-FU 400 mg/m2 iv bolus and then 600 mg/m2 iv over 22 hrs, d 1 and d2 Oxaliplatin (Eloxatin) 85 mg/m2 iv d1 Q2w x 12 cycles

SUMMARY:
This is a retrospective cost-minimization analysis study to compare the costs of treatment with EOF vs EOX regimens in patients with gastric cancer (GC) in Hong Kong. Patient baseline characteristics and cost data will be extracted from records and compared.

DETAILED DESCRIPTION:
Background

The oral chemotherapy agent Xeloda® was recently extended by the Hong Kong Hospital Authority as subsidized therapy for the treatment of colorectal cancer1. Xeloda®-based chemotherapy regimen has shown to be more cost-effective than 5-fluorouracil (5-FU) considering they had equivalent clinical efficacy in colorectal cancer treatment2,3. The total cost for 5-FU-based regimen was higher for the healthcare provider and society as a whole. Gastric cancer ranks fourth in cancer-related cause of death in the Hong Kong population4. 5-FU has known antitumor activity and has been used successfully in advanced gastric cancer (aGC) with cisplatin (FP), as well as with oxaliplatin ± epirubicin (FOLFOX4, EOF). When substituted with Xeloda®, the XP and EOX regimens have demonstrated to be noninferior in terms of progression-free survival when compared with FP and EOF, respectively5,6. In an economics evaluation done by the manufacturer for NICE submission on the use of Xeloda® for treatment of aGC, the use of XP regimen allowed a cost reduction while eliminating possible complication related to intravenous therapy7. Moreover, FOLFOX4, one of the common 5-FU-based regimens used locally, has demonstrated to produce a median overall survival of 10 months in advanced/metastatic gastric cancer patients8. An effect similar to that of EOX. Currently, there is no local data suggesting similar economic impact with Xeloda®-based regimen for gastric cancer when compared with 5-FU-based regimens. It is worthwhile to see if Xeloda®-based therapy for gastric cancer is a cost-effective alternative.

Study Objective

To compare retrospective costs of treatment with Xeloda®-based and 5-FU-based regiments in patients with advanced gastric cancer in Hong Kong.

Methods

This is a retrospective cost-minimization study to be conducted in a public hospital in Hong Kong. Sixty (60) gastric cancer patients will be identified from existing case records (30 who completed a Xeloda®-based regimen and 30 who completed a 5-FU-based regimen) in the study sites. Baseline characteristics from both groups prior to chemotherapy, including demographics, ECOG performance score, liver/renal function, metastases, and survival will be obtained. Cost data will also be extracted from patient records.

Information to be collected include cost of hospital admission and length of stay, outpatient visits, diagnostic tests and treatments, chemotherapy regimens, all other drug therapy, adverse side effect management, travel, and patient time. Baseline characteristics and costs will be compared. Descriptive statistics will be utilized and sensitivity analysis will be performed to investigate the robustness of the cost model.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were diagnosed with gastric cancer and completed either EOX or EOF chemotherapy treatment

Exclusion Criteria:

* Patients less than 18 years of age
* Patient who did not meet inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CDARS data will be accessed at respective sites to identify patients with aGC who have completed either EOX or EOF regimens.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2011-10; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Princess Margaret Hospital, Kowloon, Hong Kong

RESULTS

PARTICIPANT FLOW:
Groups:
- Epirubicin + Oxaliplatin + Capecitabine (EOX): Epirubicin + Oxaliplatin + Capecitabine (EOX) Epirubicin 50 mg/m2 iv bolus d1 q3w x 8 cycles Oxaliplatin (Eloxatin) 130 mg/m2 iv over 2 hours d1 q3w x 8 cycles Capecitabine (Xeloda) 625 mg/m2 po bid x 6 months
Period: Overall Study
Arm/Group | Epirubicin + Oxaliplatin + Capecitabine (EOX) | FOLFOX4
Started | 45 | 13
Completed | 45 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Epirubicin + Oxaliplatin + Capecitabine (EOX) | FOLFOX4 | Total
Number analyzed (Participants) | 45 | 13 | 58
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 12 | 52
  >=65 years | 5 | 1 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (10) | 56.5 (13.3) | 56.5 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 5 | 24
  Male | 26 | 8 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 45 | 13 | 58
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Hong Kong | 45 | 13 | 58
ECOG Performance Scores < 2 [Count of Participants; unit: Participants] | 42 | 10 | 52
ECOG Performance Score >= 2 [Count of Participants; unit: Participants] | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Expected and Unexpected Provider Costs
Description: Expected and unexpected provider costs (chemotherapy, hospital stay, lab tests, clinic visits, AE management, other drug costs). The costs for healthcare resources usage, including hospital visits and laboratory investigations, were valued according to the Hong Kong Government Gazette 2003, which is the most updated version of official source for costs of public hospital services.
Time Frame: At the completion of respective chemotherapy regimen, up to 6 months
Measure: Mean (Standard Deviation); unit: HK$
Groups:
- EOX (Epirubicin, Oxaliplatin, Xeloda®- Capecitabine): It consists of an intravenous bolus injection of epirubicin 50 mg/m2 and an intravenous infusion of oxaliplatin 130 mg/m2 over 2 hours on day 1 of every 3 week cycles, together with oral capecitabine tablets 625 mg/m2 twice daily for six months.
- FOLFOX4 (5-fluorouracil (5-FU), Leucovorin, Oxaliplatin): It consists of an intravenous infusion of oxaliplatin 85 mg/m2 over 2 hours on day 1, and an intravenous infusion of folinic acid (leucovorin) 200 mg/m2 over 2 hours on days 1 and 2. This is followed by an intravenous bolus injection of 5-FU 400 mg/m2 and then continuous intravenous infusion of 5-FU 600 mg/m2 over 22 hours every 2 weeks.
Arm/Group | EOX (Epirubicin, Oxaliplatin, Xeloda®- Capecitabine) | FOLFOX4 (5-fluorouracil (5-FU), Leucovorin, Oxaliplatin)
Number analyzed (Participants) | 45 | 13
HK$
  Expected Medication Cost | 2264.1 (354.5) | 522 (104.5)
  Expected Laboratory Tests | 1135.7 (294.3) | 846 (200.2)
  Expected Day ward/inpatient visits | 600 (0) | 9900 (0)
  Expected X rays & Scans | 760.3 (361.2) | 846.9 (367.6)
  Expected Outpatient visits | 1094.3 (263) | 864.8 (163.2)
  Unexpected Medication Cost | 116.2 (255.4) | 112.3 (169.9)
  Unexpected Emergency unit visit | 39.5 (74.3) | 85.8 (109.6)
  Unexpected Hosptial Bed-days | 1531.4 (4607.9) | 2830.5 (4358.6)
  Unexpected Laboratory Tests | 297 (256.9) | 497.5 (470.5)
  Unexpected X rays & Scans | 211.8 (520.1) | 315.6 (785.5)
  Unexpected Outpatient visits | 344.1 (251.3) | 404.7 (433.3)
  Total Unexpected Cost/cycle | 2540.1 (5064.4) | 4246.4 (4875.1)
  Total Unexpected Cost/patient | 13434.0 (26785.2) | 33546.6 (38250.8)
  Total Cost/patient | 44397.1 (27105.7) | 135387.9 (39084.0)

2. Secondary Outcome: Expected and Unexpected Societal Costs
Description: Expected and unexpected societal costs (patient time, travel)
Time Frame: At the completion of respective chemotherapy regimen, up to 6 months
Measure: Mean (Standard Deviation); unit: HK$
Groups:
- Epirubicin + Oxaliplatin + Capecitabine (EOX) Group: Epirubicin + Oxaliplatin + Capecitabine (EOX) Epirubicin 50 mg/m2 iv bolus d1 q3w x 8 cycles Oxaliplatin (Eloxatin) 130 mg/m2 iv over 2 hours d1 q3w x 8 cycles Capecitabine (Xeloda) 625 mg/m2 po bid x 6 months
Arm/Group | Epirubicin + Oxaliplatin + Capecitabine (EOX) Group | FOLFOX4
Number analyzed (Participants) | 45 | 13
HK$
  Expected Patient Time Cost | 544 (154.4) | 1013.1 (471.4)
  Expected Patient Travel Cost | 402.7 (290.5) | 236.6 (118.5)
  Expected Patient Treatment Cost | 3097.1 (468.1) | 2322.5 (267.7)
  Total Expected Cost/Cycle | 4043.7 (707.7) | 3572.2 (354.9)
  Total Expected Cost/Patient | 21386.7 (3742.7) | 28220.4 (2784.8)
  Unexpected Patient Time Cost | 323.3 (489.2) | 306.3 (400.3)
  Unexpected Patient Travel Cost | 106.2 (110.7) | 69.5 (63.5)
  Unexpected Patient Treatment Cost | 84.6 (141.1) | 134.7 (137.6)
  Total Unexpected Cost/Cycle | 514.1 (645) | 510.5 (538.1)
  Total Cost/Patient | 2719.3 (3517) | 4033 (4221.7)

ADVERSE EVENTS:
Arm/Group | EOX (Epirubicin, Oxaliplatin, Xeloda®- Capecitabine) | FOLFOX4 (5-fluorouracil (5-FU), Leucovorin, Oxaliplatin)
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/13
Other Adverse Events (participants affected / at risk) | 22/45 | 7/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EOX (Epirubicin, Oxaliplatin, Xeloda®- Capecitabine) (N=45) | FOLFOX4 (5-fluorouracil (5-FU), Leucovorin, Oxaliplatin) (N=13)
Nausea and Vomiting (Gastrointestinal disorders) | 22 (30) | 7 (14) — For both groups, nausea and vomiting were the most commonly associated adverse events; hence the most frequently used medications were anti-emetic drugs.

LIMITATIONS AND CAVEATS:
1. A total of 58 subjects were identified with only thirteen in the FOLFOX4 arm. The two groups were then arranged for comparison in an approximate 3:1 ratio (45 EOX and 13 FOLFOX4). More patients seem to have chosen EOX over FOLFOX4 to avoid the inpatient stay for the prolonged administration of FOLFOX4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No